CLINICAL TRIAL: NCT06027268
Title: ToPCourT: A Phase II Trial of Trilaciclib, Pembrolizumab, Gemcitabine and Carboplatin in Locally Advanced Unresectable or Metastatic Triple-Negative Breast Cancer (TNBC)
Brief Title: Phase II Trial of Trilaciclib, Pembrolizumab, Gemcitabine and Carboplatin in Metastatic Triple-Negative Breast Cancer
Acronym: ToPCourT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); G1 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00095334; LCI-BRE-MTN-TPGC-001 (Other: Atrium Health)
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Triple-Negative Breast Cancer
Keywords: Breast-Female; Breast-Male; Triple-Negative Breast Cancer; Metastatic; Locally advanced unresectable
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Neoplasm Metastasis | interventions — trilaciclib; pembrolizumab; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Trilaciclib, Pembrolizumab, Gemcitabine, and Carboplatin (Experimental): Trilaciclib is an agent that helps protect the bone marrow from the side effects of chemotherapy. It is given as an intravenous (IV) infusion over 30 minutes prior to gemcitabine and carboplatin. Gemcitabine is given IV over 30 minutes. Carboplatin is given over 30 minutes. Trilaciclib, gemcitabine and carboplatin are given on Days 1 and 8 every 21 days. Pembrolizumab is given IV over 30 minutes on Day 1 every 21 days.
  Interventions: Drug: Trilaciclib; Drug: Pembrolizumab; Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Trilaciclib — IV infusion Day 1 and Day 8 every 21 days, at dose of 240 mg/m2
  Other Names: COSELA
Drug: Pembrolizumab — IV infusion Day 1 every 21 days, at dose of 200 mg
  Other Names: KEYTRUDA
Drug: Gemcitabine — IV infusion Day 1 and Day 8 every 21 days, at dose 1000 mg/m2
  Other Names: Gemzar
Drug: Carboplatin — IV infusion Day 1 and Day 8 every 21 days, at dose area under curve (AUC) 2 (maximum of 300 mg)

SUMMARY:
The goal of this phase II study is to test the combination of trilaciclib, pembrolizumab, gemcitabine, and carboplatin in locally advanced unresectable or metastatic triple-negative breast cancer.

The main questions it aims to answer are:

* to evaluate the anti-cancer efficacy (assess how well it works)
* to evaluate the safety and tolerability (how well the body can handle the treatment) of this combination of anti-cancer therapy

DETAILED DESCRIPTION:
This is an open label, single-arm, phase II trial designed to evaluate the efficacy of trilaciclib, pembrolizumab, gemcitabine and carboplatin in participants with locally advanced unresectable or metastatic triple-negative breast cancer. Pembrolizumab will be given for a maximum of 2 years. Eligible participants will receive the study treatment until disease progression, unacceptable toxicity, or withdrawal for any reason. A tumor biopsy will be collected from participants in which it can be safely obtained before the first dose of treatment, prior to Cycle 3 Day 1, and at the time of disease progression (optional). Blood specimens for correlative studies will be collected pre-treatment Cycle 1 Day 1, prior to treatment Cycle 2 Day 1, prior to treatment Cycle 3 Day 1, 3 months after the start of study treatment, and 6 months after the start of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information signed by the patient
2. Male or female with locally advanced unresectable or metastatic TNBC
3. Age ≥ 18 years at the time of consent
4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1 evaluated within 28 days prior to day 1 of study treatment
5. Histological or cytological confirmation of estrogen negative and progesterone negative tumor, defined as < 10% staining on immunohistochemistry (IHC) and human epidermal growth factor receptor type 2 (HER2)-negative, defined as HER 2 IHC 0 or 1+ or IHC 2+ with no amplification. Patients may be enrolled regardless of their PD-L1 (programmed death ligand-1) status.
6. Measurable disease according to response evaluation criteria in solid tumors
7. Demonstrate adequate organ function
8. Female patients: All females of childbearing potential must have a negative serum β-human chorionic gonadotropin (hCG) test result at Screening and negative serum or urine pregnancy test results within 72 hours prior to day 1 of study treatment.
9. Subject agrees to use contraception
10. As determined by the enrolling physician, the ability of the subject to understand and comply with study procedures for the entire length of the study
11. Tumor tissue: Willing to provide tumor tissue for research purposes
12. Subject has a life expectancy of ≥ 12 weeks

Exclusion Criteria:

1. More than 3 prior lines of chemotherapy for locally advanced unresectable or triple-negative metastatic disease
2. Prior therapy with the concurrent combination of gemcitabine and carboplatin in the metastatic setting
3. Active, symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis or CNS metastases that are progressing on screening magnetic resonance imaging (MRI) brain.
4. Prior systemic anti-cancer therapy within 3 weeks, prior stereotactic radiotherapy within 1 week, and radiation within 2 weeks of day 1 of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation to non-CNS disease.
5. Major surgery, defined by the investigator's discretion, within 3 weeks of day 1 of study treatment
6. Not recovered from all reversible acute toxic effects of prior therapy, including non-hematologic toxicities related to prior systemic therapy to ≤ Grade 1. Participants with less than Grade 2 neuropathy or alopecia of any grade are an exception
7. Active infection requiring systemic therapy
8. Pregnant or breastfeeding
9. Participants previously diagnosed with an additional malignancy must be disease-free for at least five years prior to enrollment. Exceptions include basal cell or squamous cell skin cancer and in situ cervical or bladder cancer.
10. Treatment with any investigational drug within 30 days or at least 5 half-lives, whichever is longer, prior to day 1 of study treatment
11. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled symptomatic congestive heart failure (Class III or IV as defined by the New York Heart Association (NYHA) functional classification system), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations/substance abuse that would limit compliance with study requirements as determined by the investigator
12. Known history of stroke or cerebrovascular event within 6 months prior to the day 1 of study treatment
13. Known hypersensitivity to carboplatin or other platinum-containing compounds, gemcitabine, mannitol, or pembrolizumab
14. History of non-infectious interstitial lung disease (ILD)/pneumonitis that required steroids or current ILD/ pneumonitis.
15. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs) prior to day 1 of study treatment. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed
16. Prior hematopoietic stem cell or bone marrow transplant or allogenic tissue/solid organ transplant
17. Has a known history of Human Immunodeficiency Virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
18. Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive).
19. Has known active hepatitis C (e.g., hepatitis C virus (HCV) ribonucleic acid (RNA) [qualitative] is detected).
20. Receipt of a live, attenuated vaccine within 30 days prior to day 1 of study treatment or anticipation that such a live, attenuated vaccine will be required during the study treatment period. Administration of killed vaccines is allowed. Exception: Monkeypox vaccine may be given if there are at least 3 days between the vaccine and initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Objective Response | 6 months (initiation of protocol directed therapy until either a partial response is achieved or treatment discontinuation)
  Objective according to RECIST v1.1 criteria

SECONDARY OUTCOMES:
Progression-free survival | 1 year (initiation of protocol directed therapy until documented disease progression, death, or end of follow-up period)
  Time to disease progression per RECIST v1.1 criteria or death
Duration of response | 1 year (time from first disease assessment that shows a PR or complete response (CR) until documented disease progression, death, or end of follow-up period)
  Duration of response will be calculated only for subjects who achieve an objective response according to RECIST v1.1 criteria (a CR or PR). Disease progression will be objectively determined as per RECIST 1.1 criteria or progression can be subjective as determined by the Investigator.
Overall survival | 1 year (initiation of protocol directed therapy until documented death, or end of follow-up period])
  Time to date of death due to any cause while on study

OTHER OUTCOMES:
Adverse Events | 30 days (initiation of protocol directed therapy until 30 days after last dose, or removal from study while on treatment)
  Trilaciclib, pembrolizumab, gemcitabine, and carboplatin treatment administration AEs while on study therapy
Serious Adverse Events | 30 days (initiation of protocol directed therapy until 30 days after last dose, or removal from study while on treatment)
  Trilaciclib, pembrolizumab, gemcitabine, and carboplatin treatment administration SAEs while on study therapy
Adverse Event Related Dose Delays | 30 days (initiation of protocol directed therapy until 30 days after last dose, or removal from study while on treatment)
  Trilaciclib, pembrolizumab, gemcitabine, and carboplatin treatment administration AE-related dose delays while on study therapy
Dose Reductions | 30 days (initiation of protocol directed therapy until 30 days after last dose, or removal from study while on treatment)
  Trilaciclib, pembrolizumab, gemcitabine, and carboplatin treatment administration dose reductions while on study therapy
Treatment Discontinuation | 30 days (initiation of protocol directed therapy until 30 days after last dose, or removal from study while on treatment)
  Trilaciclib, pembrolizumab, gemcitabine, and carboplatin treatment administration treatment discontinuation while on study therapy
Deaths | 30 days (initiation of protocol directed therapy until 30 days after last dose, or removal from study while on treatment)
  Trilaciclib, pembrolizumab, gemcitabine, and carboplatin treatment administration deaths while on study therapy

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Tan, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tan AR, Wright GS, Thummala AR, Danso MA, Popovic L, Pluard TJ, Han HS, Vojnovic Z, Vasev N, Ma L, Richards DA, Wilks ST, Milenkovic D, Yang Z, Antal JM, Morris SR, O'Shaughnessy J. Trilaciclib plus chemotherapy versus chemotherapy alone in patients with metastatic triple-negative breast cancer: a multicentre, randomised, open-label, phase 2 trial. Lancet Oncol. 2019 Nov;20(11):1587-1601. doi: 10.1016/S1470-2045(19)30616-3. Epub 2019 Sep 28. PMID 31575503
- [Background] Tan AR, Wright GS, Thummala AR, Danso MA, Popovic L, Pluard TJ, Han HS, Vojnovic Z, Vasev N, Ma L, Richards DA, Wilks ST, Milenkovic D, Xiao J, Sorrentino J, Horton J, O'Shaughnessy J. Trilaciclib Prior to Chemotherapy in Patients with Metastatic Triple-Negative Breast Cancer: Final Efficacy and Subgroup Analysis from a Randomized Phase II Study. Clin Cancer Res. 2022 Feb 15;28(4):629-636. doi: 10.1158/1078-0432.CCR-21-2272. PMID 34887261
- [Background] Tan AR, O'Shaughnessy J, Cao S, Ahn S, Yi JS. Investigating potential immune mechanisms of trilaciclib administered prior to chemotherapy in patients with metastatic triple-negative breast cancer. Breast Cancer Res Treat. 2023 Sep;201(2):307-316. doi: 10.1007/s10549-023-07009-8. Epub 2023 Jul 7. PMID 37418031